CLINICAL TRIAL: NCT02825940
Title: A Phase I, Open-Label Study to Assess the Pharmacokinetics, Efficacy, and Safety of Atezolizumab Administered Intravenously as a Single Agent or in Combination With Chemotherapy in Chinese Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess the Pharmacokinetics, Efficacy, and Safety of Atezolizumab Administered Intravenously (IV) as a Single Agent or in Combination With Chemotherapy in Chinese Participants With Locally Advanced or Metastatic Solid Tumors
Acronym: IMYO29233
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO29233
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Gemcitabine; Cisplatin

ARMS (2):
- Atezolizumab Monotherapy: PK and Extension Phases (Experimental): Participants during the PK and extension phases of the study will receive atezolizumab alone at a dose of 1200 milligrams (mg) IV every 3 weeks (q3w) (in 21-day cycles) continuously until loss of clinical benefit, disease progression, unacceptable toxicity, participant or physician decision to discontinue, or death. Study treatment may continue beyond disease progression based on the investigator's discretion.
  Interventions: Drug: Atezolizumab
- Atezolizumab and Chemotherapy: Extension Phase (Experimental): Participants during the extension phase of the study will receive atezolizumab at a dose of 1200 mg IV on Day 1 in combination with gemcitabine at a dose of 1250 milligrams per square meter (mg/m^2) on Days 1 and 8 and cisplatin at a dose of 75 mg/m^2 on Day 1 (four or six 21-day cycles at the discretion of the investigator), followed by atezolizumab as a single agent at a dose of 1200 mg IV q3w on Day 1 of a 21-day cycle) as maintenance treatment continuously until loss of clinical benefit, disease progression, unacceptable toxicity, participant or physician decision to discontinue, or death. Study treatment may continue beyond disease progression based on the investigator's discretion.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg IV q3w (in 21-day cycles), except for participants with NSCLC who will be administered atezolizumab at a dose of 1200 mg IV on Day 1.
  Other Names: MPDL3280A; RO5541267
Drug: Gemcitabine — Gemcitabine will be administered to participants with NSCLC at a dose of 1250 mg/m^2 on Days 1 and 8.
  Arms: Atezolizumab and Chemotherapy: Extension Phase
Drug: Cisplatin — Cisplatin will be administered to participants with NSCLC at a dose of 75 mg/m^2 on Day 1.
  Arms: Atezolizumab and Chemotherapy: Extension Phase

SUMMARY:
This Phase I, open-label, multicenter study will evaluate the pharmacokinetics, safety, and preliminary anti-tumor activity of atezolizumab as monotherapy in Chinese participants with locally advanced or metastatic gastric cancer, nasopharyngeal cancer, esophageal cancer, and hepatocellular carcinoma (HCC) that are refractory to standard therapeutic modalities and for whom no further standard therapy is available or who have refused standard therapy; and the safety and preliminary anti-tumor activity of atezolizumab in combination with gemcitabine and cisplatin in Chinese participants with Stage IV, treatment-naive non-small cell lung cancer (NSCLC). The study will consist of a pharmacokinetic (PK) phase and an extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, incurable or metastatic solid tumor that is advanced (non-resectable) or recurrent and progressing since the last the anti-tumor therapy and for which no recognized standard curative therapy exists or who have refused the standard therapy
* Adequate hematologic and end organ function
* Measurable disease per RECIST v1.1 or mRECIST
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Women who are not postmenopausal (greater than or equal to (>=) 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment
* A representative formalin-fixed paraffin-embedded (FFPE) tumor specimen in paraffin block (preferred) or 15 or more unstained, freshly cut, serial sections (on slides) from an FFPE tumor specimen is required for participation in this study. This specimen must be accompanied by the pathology report
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1% per year during the treatment period and for at least 90 days 5 months after the last dose of atezolizumab, or 6 months after the last dose of cisplatin or gemcitabine, whichever is longer, if combined. Women must refrain from donating eggs during this same period
* For men in the NSCLC cohort only: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm
* For participants in the NSCLC Cohort: Histologically or cytologically confirmed Stage IV NSCLC (per the Union Internationale contre le Cancer/American Joint Committee on Cancer staging system)
* For participants in the NSCLC Cohort: No prior chemotherapy for Stage IV NSCLC
* For participants in the NSCLC Cohort: Participants who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from enrollment since the last chemotherapy, radiotherapy, or chemoradiotherapy cycle

Exclusion Criteria:

* Pregnant or lactating
* Any approved anti-cancer therapy, including chemotherapy, targeted therapy or hormonal therapy less than (<) 5 half-lives prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Uncontrolled hypercalcemia (greater than (>) 1.5 millimoles per liter (mmol/L) ionized calcium or calcium >12 milligram per deciliter (mg/dL) or corrected serum calcium greater than the upper limit of normal) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease, uncontrolled major seizure disorder, or superior vena cava syndrome
* Participants with acute leukemia, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
* Symptomatic, actively progressing, or untreated central nervous system metastases as determined by computed tomography or magnetic resonance imaging evaluation during screening and prior radiographic assessments
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Participants with prior allogenic stem cell or solid organ transplantation
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participant at high risk from treatment complications
* Positive test for HIV
* Participants with active hepatitis B infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C infection (for the non-HCC cohorts only)
* For participants in the NSCLC Cohort: Known tumor programmed death-ligand 1 (PD-L1) expression status as determined by an immunohistochemistry assay during participation in other clinical studies (e.g., participants whose PD-L1 expression status was determined during screening for entry into a study with anti-programmed death 1 or anti-PD-L1 antibodies but were not eligible are excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Atezolizumab | Pre-dose (0 hours [h]), 0.5h post-dose (PtD) at Day (D) 1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Minimum Observed Plasma Concentration (Cmin) of Atezolizumab | Pre-dose (0h), 0.5h PtD at D1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Accumulation Ratio (R) of Atezolizumab Based on Concentrations After the First Dose and at Steady State | Pre-dose (0h), 0.5h PtD at D 1; D2, 4, 8, 15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Area Under the Plasma Concentration-Time Curve (AUC) of Atezolizumab (PK phase only) | Pre-dose (0h), 0.5h PtD at D 1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Systemic Clearance (CL) of Atezolizumab (PK phase only) | Pre-dose (0h), 0.5h PtD at D1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Volume of Distribution at Steady State (Vss) of Atezolizumab (PK phase only) | Pre-dose (0h), 0.5h PtD at D1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Terminal Half-Life (t1/2) of Atezolizumab (PK phase only) | Pre-dose (0h), 0.5h PtD at D1; D2,4,8,15 of C1; pre-dose (-2h), 0.5h PtD at D1 of C2,3,4,8,12,16, thereafter every eight cycles until treatment discontinuation or 120 days after last dose (maximum up to 3 years)
Objective Response (OR), Defined as a Complete Response (CR) or Partial Response (PR) on Two Consecutive Occasions >/= 4 Weeks Apart, as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | From the first occurrence of a PR or CR through the end of study (maximum up to 3 years)

SECONDARY OUTCOMES:
Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1 | From the first occurrence of a documented OR to the first occurrence of disease progression, whichever occurs first (maximum up to 3 years)
Time to Progression (TTP) (HCC Cohort) as Determined by the Investigator According to RECIST v1.1 | From the first dose of atezolizumab (Day 1) to the first occurrence of disease progression (maximum up to 3 years)
Progression-free Survival (PFS) as Determined by the Investigator According to RECIST v1.1 | From the first dose of atezolizumab (Day 1) to the first occurrence of disease progression or death, whichever comes first (maximum up to 3 years)
Overall survival (OS) | From the first dose of atezolizumab (Day 1) to death from any cause (maximum up to 3 years)
OS at 6 Months and 1 Year | 6 Months; 1 Year
Percentage of Participants with Adverse Events (AE) | From baseline through the end of study (maximum up to 3 years)
Percentage of Participants with Anti-Therapeutic Antibodies (ATA) to Atezolizumab | From first dose of atezolizumab (Day 1) through the end of study (maximum up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Cancer Center, Sun Yat-sen University of Medical Sciences; Department of Medical Oncology, Guangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai